CLINICAL TRIAL: NCT01984515
Title: Increasing Engagement in Evidence-Based PTSD Therapy for Primary Care Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRP 13-204
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Results first posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-11

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Post-traumatic Stress Disorder; Evidence-Based Psychotherapy; Treatment Engagement; Cognitive Behavioral Therapy; Implementation Science
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Team Red Primary Care (Experimental): Eligible patients will receive the Referral Management System in primary care
  Interventions: Behavioral: Referral Management System

INTERVENTIONS:
Behavioral: Referral Management System — Referral Management System (RMS) will address patient-level barriers with the delivery of a 1-session cognitive behavioral therapy (CBT) intervention to identify and change treatment seeking beliefs that serve as an barrier to treatment engagement, including specific negative beliefs about EBP (e.g., "talking about past trauma will be too difficult for me"). RMS will address system-level barriers by tracking the progress of RMS referrals and contacting Veterans who have not followed thought on their chosen referral options. Primary Care staff will also be trained with simple scripts on how to address PTSD symptoms and make appropriate referrals based on VA/DoD Clinical Practice Guidelines for PTSD.

SUMMARY:
The purpose of this study is to implement an evidence-based Referral Management System that will address patient and system-level barriers to the uptake of evidence-based psychotherapy for PTSD by Veterans Affairs primary care patients.

DETAILED DESCRIPTION:
Within the Veteran's Health Administration (VHA), primary care (PC) patients with PTSD have low rates of engagement in evidence-based psychotherapy (EBP) for PTSD. Low engagement rates are due to a variety of patient-level (e.g., belief that treatment will not be helpful, stigma) and system-level barriers (e.g., lack of tracking of referral process, knowledge gaps on how to manage PTSD). We propose to conduct a pilot hybrid effectiveness- implementation study to implement an evidence-based Referral Management System (RMS) that will address patient and system-level barriers to the uptake of EBP for PTSD by VHA primary care patients. RMS will address patient-level barriers with the delivery of a 1-session cognitive behavioral therapy (CBT) intervention to identify and change treatment seeking beliefs that serve as an barrier to treatment engagement, including specific negative beliefs about EBP (e.g., talking about past trauma will be too difficult for me"). This CBT intervention has been previously found to be effective for increasing treatment engagement with Veterans with PTSD. Depending on Veteran preference, it will be delivered by the PC-MHI provider within the PC clinic or a Behavioral Health Lab (BHL) care manager by phone. RMS will be initiated by PACT staff and will address system-level barriers by having a BHL technician track the progress of RMS referrals and contact Veterans who have not followed thought on their chosen referral options. PACT staff will also be trained with simple scripts on how to address PTSD symptoms and make appropriate referrals based on VA/DoD Clinical Practice Guidelines for PTSD. Our aims, implementation strategy, data collection, and analyses will be guided by established strategies. The Consolidated Framework for Implementation Research (CFIR) will identify organization variables. RE-AIM will investigate program uptake and patient/ system-level impact. An Implementation Mapping approach will guide our implementation strategy. We propose to conduct this study in 3 phases. Phase 1 includes interviews with PC and MH leadership about the relevance of CFIR constructs to RMS implementation and a meeting with PACT staff to train them on RMS and gather their input on how RMS should be adapted to their clinic. A PC medical provider will serve as a clinical champion who is knowledgeable, communicative, and a leader in promoting RMS among his/her peers. Phase 2 consists of implementing RMS for 6 months in one Syracuse PC clinic and then measuring RE-AIM outcomes. Some RE-AIM outcomes compared participants who received RMS to those who did not receive RMS in a historical control group. Phase 3 involves meeting with PACT and MH Leadership and PACT staff to share a formal report of study results and gather information about potential barriers and facilitators to long-term maintenance and future expansion of RMS within the CFIR framework. An expert national stakeholder panel will also be convened to guide development of a SDP that will investigate multi-VISN implementation.

Our long-term aim of this line of research is to increase implementation of evidence-based psychotherapy for PTSD by getting more primary care patients with PTSD to engage in treatment.

Our Specific Aims for this Rapid Response Project are to:

1. Assess and improve the feasibility of implementing RMS in PC-MHI/PACT settings

1A. Diagnose organizational and staff-level barriers and facilitators to implementing RMS.

1B. Adapt RMS for the local context based on information gathered about barriers and facilitators.

2. Evaluate initial impact of implementing RMS in PC-MHI/PACT settings. Assess impact of RMS on RE-AIM measures of Reach, Efficacy/Effectiveness, Adoption, Implementation and Maintenance 3. Refine implementation strategy based on study findings for planned efforts to spread RMS to additional VISNs in a QUERI Phase 2 Service-Directed Project (SDP) to follow.

ELIGIBILITY:
Inclusion Criteria:

* Team Red primary care patients,
* have a score of at least 44 on PCL-S and
* able to give informed consent.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Possemato, PhD, Principal Investigator — Syracuse VA Medical Center, Syracuse, NY
Locations (1):
- Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Team Red Primary Care
Started | 59
Received CBT Session | 40
Completed | 40
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | Team Red Primary Care
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — self-report
  Participants
    Hispanic or Latino | 3
    Not Hispanic or Latino | 37
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Engagement in Evidence-based Psychotherapy for PTSD
Description: Engagement will be assessed by how many patients attend at least 2 sessions of an evidence-based psychotherapy for PTSD and how many complete treatment. Completion is defined as 8 sessions.
Time Frame: From initiation of the Referral Management System to 6 months after initiation
Measure: Number; unit: participants
Arm/Group | Team Red Primary Care
Number analyzed (Participants) | 40
participants | 40

2. Secondary Outcome: PTSD Checklist-Specific
Description: Measures the 17 symptoms of PTSD according to the DSM-IV. Scale for each item ranges from 1-5. Total scale score ranges from 17-85. 17 represents no PTSD symptoms and 85 represented the most severe PTSD symptoms.
Time Frame: Referral Management Initiation, 1 month post initiation, 3 months post initiation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Team Red Primary Care
Number analyzed (Participants) | 40
units on a scale
  RMS initiation | 64 (10)
  1 month post initiation | 59 (9)
  3 months post initiation | 59 (12)

3. Secondary Outcome: Patient Health Questionnaire-9 Item
Description: 9 symptoms of depression are measured on a 0-3 scale. Total scale range is 0-27, with higher scores indicating worse depression.
Time Frame: Referral Management Initiation, 1 month post initiation, 3 months post initiation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Team Red Primary Care
Number analyzed (Participants) | 40
units on a scale
  RMS initiation | 16 (5)
  1 month post RMS initiation | 14 (4)
  3 months post RMS initiation | 14 (5)

ADVERSE EVENTS:
Arm/Group | Team Red Primary Care
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes